CLINICAL TRIAL: NCT03301883
Title: A Phase IV, Multicenter, Single-Arm, Open-Label Study to Assess the Efficacy and Safety of Tocilizumab in Chinese Patients With Systemic Juvenile Idiopathic Arthritis
Brief Title: A Study of Tocilizumab in Chinese Participants With Systemic Juvenile Idiopathic Arthritis (sJIA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YA39368
Record Dates: First submitted 2017-09-21; First posted 2017-10-04 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — tocilizumab; Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tocilizumab (Experimental): Participants weighing greater than or equal to (>/=) 30 kilograms (kg) will receive tocilizumab 8 milligrams per kilogram (mg/kg) intravenous (IV) infusion every 2 weeks (Q2W), and participants weighing less than (<) 30 kg will receive tocilizumab 12 mg/kg IV infusion Q2W for 52 weeks. After Week 12, the dose of tocilizumab can be adjusted for non-transient changes in body weight (shifting from <30 to >/=30 kg) over a minimum of three consecutive dosing visits. MTX, NSAIDs, and oral corticosteroids (CSs) are permitted but not required during the study.
  Interventions: Drug: Tocilizumab; Drug: NSAIDs; Drug: CSs; Drug: MTX

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab will be administered as per the schedule specified in the arm description.
  Other Names: RO4877533
Drug: NSAIDs — Participants may receive NSAIDs up to the maximum recommended stable daily dose. Study protocol does not enforce any particular NSAID.
Drug: CSs — Participants may receive CSs at a stable dose of 30 milligrams per day (mg/day) or 0.5 milligrams per kilogram per day (mg/kg/day), whichever is less. Study protocol does not enforce any particular CS.
Drug: MTX — Participants may receive MTX at a stable dose of less than or equal to (</=) 20 milligrams per square meter (mg/m^2).

SUMMARY:
This Phase IV, multicenter, single-arm, open-label study will evaluate the efficacy and safety of tocilizumab in Chinese participants with sJIA with persistent activity and an inadequate response to non-steroidal anti-inflammatory drugs (NSAIDs) and steroid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants meeting International League of Associations for Rheumatology (ILAR) classification for sJIA
* Greater than (>) 6 months of documented persistent sJIA activity prior to screening
* Active disease
* hsCRP >4.3 milligrams per liter (mg/L) or 0.43 milligrams per deciliter (mg/dL)
* Participant who has recovered from any symptomatic serositis for at least 30 days prior to the screening visit, and requires a dose of CSs at baseline of </=30 mg/day or </=0.5 mg/kg/day, whichever is less
* Participants meeting one of the following: Participant who is not receiving MTX or discontinued MTX >/=4 weeks prior to baseline visit; participant who has been taking MTX >/=12 weeks immediately prior to the baseline visit and on a stable dose of </=20 mg/m^2 for >/=8 weeks prior to the baseline visit, together with either folic acid or folinic acid according to local standard of care
* Participant who was never treated with biologics or, if was previously treated with biologics, discontinued etanercept (or Yisaipu, Qiangke, or Anbainuo) >/=2 weeks, infliximab or adalimumab >/=8 weeks, anakinra >/=1 week, or abatacept >/=12 weeks prior to the baseline visit
* Participant who is not currently receiving oral CSs, or is taking oral CSs at a stable dose for >/=2 weeks prior to the baseline visit at </=30 mg/day or </=0.5 mg/kg/day, whichever is less
* Participant who is not taking NSAIDs, or taking </=1 type of NSAID at a stable dose for >/=2 weeks prior to the baseline visit and is less than or equal to the maximum recommended daily dose

Exclusion Criteria:

* Wheelchair bound or bedridden participant
* Any other autoimmune, rheumatic disease, or overlap syndrome other than sJIA
* Participant who is not fully recovered from recent surgery or <6 weeks since surgery at the time of screening visit; or planned surgery during the initial 12 weeks of the study
* Lack of peripheral venous access
* Any significant concurrent medical or surgical condition that would jeopardize the participant's safety or ability to complete the trial
* Evidence of serious uncontrolled concomitant diseases
* Asthma for which the participant has required the use of oral or parenteral CSs for >/=2 weeks within 6 months prior to the baseline visit
* Known human immunodeficiency (HIV) infection or other acquired forms of immune compromise or congenital conditions characterized by a compromised immune system
* Any active acute, subacute, chronic, or recurrent bacterial, mycobacterial, viral, or systemic fungal infection or opportunistic infection
* Any major episode of infection requiring hospitalization or treatment during screening, treatment with IV antibiotics completing within 4 weeks of the screening visit, or oral antibiotics completing within 2 weeks of the screening visit
* History of atypical tuberculosis (TB)
* Active TB requiring treatment within 2 years prior to screening visit
* Positive purified protein derivative (PPD) or T-spot test (interferon-gamma [IFN-γ]-based test) at screen
* Positive for latent TB
* History of reactivation or new onset of a systemic infection such as herpes zoster or Epstein-Barr virus (EBV) within 2 months of the screening visit
* Hepatitis B surface antigen (Ag)- or hepatitis C antibody (Ab)-positive
* History of macrophage activation syndrome (MAS) within 3 months prior to the screening visit
* Evidence of active malignant disease or diagnosed malignancies
* Uncontrolled diabetes mellitus
* Previous treatment with tocilizumab
* Intra-articular, intramuscular, IV, or long-acting CSs administration within 28 days prior to the baseline visit
* Treatment with non-biologic disease-modifying antirheumatic drugs (DMARDs; other than MTX) within 6 weeks prior to the baseline visit
* Treatment with leflunomide that was not followed by standardized cholestyramine washout and documented to be below the limit of detection prior to the baseline visit
* Treatment with cyclophosphamide, etoposide (VP16) and statins within 90 days prior to the baseline visit
* Treatment with growth hormone and androgens within 4 weeks prior to the baseline visit
* Administration of IV immunoglobulin within 28 days prior to the baseline visit
* Treatment with any cell-depleting therapies
* Stem cell transplant at any time
* Participant who has received live or attenuated vaccines within 4 weeks prior to the baseline visit, or intending to receive while on study drug or 3 months following the last dose of study drug

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Juvenile Idiopathic Arthritis (JIA) American College of Rheumatology (ACR) 30 (JIA ACR30) Response With Absence of Fever, at Week 12 | Week 12

SECONDARY OUTCOMES:
Percentage of Participants Achieving JIA ACR30 Response With Absence of Fever, at Week 52 | Week 52
Percentage of Participants With 30 Percent (%), 50%, 70%, and 90% Improvement From Baseline in JIA Core Set Parameters | Baseline, Weeks 12, 24, and 52
Percentage of Participants With Inactive Disease Assessed According to Criteria for Inactive Disease and Clinical Remission of sJIA (Wallace et. al. 2011 Criteria) | Weeks 24 and 52
Percentage of Participants With Clinical Remission Assessed According to Criteria for Inactive Disease and Clinical Remission of sJIA (Wallace et. al. 2011 Criteria) | Week 52
Percentage of Participants With an Elevated High-Sensitivity C-Reactive Protein (hsCRP) Levels at Baseline Who Have Normal hsCRP Levels at Weeks 12, 24, and 52 | Baseline, Weeks 12, 24, and 52
Mean Glucocorticoid Dose | Baseline up to Week 52
Mean Methotrexate (MTX) Dose | Baseline up to Week 52
Change From Baseline in Glucocorticoid Dose | From Baseline to Week 52
Change From Baseline in MTX Dose | From Baseline to Week 52
Pain Visual Analog Scale (VAS) Score | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Change From Baseline in Pain VAS Score | Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Percentage of Participants Who Discontinue Permitted Concomitant Medication for sJIA | Baseline up to Week 52
Percentage of Participants With Adverse Events (AEs) | Baseline up to end of study (up to Week 60)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- China (10):
  - Capital Institute of Pediatrics, Beijing
  - Beijing Children's Hospital, Capital Medical University; rheumatism, Beijing
  - The First Hospital of Jilin University, Changchun
  - Children's Hospital Chongqing Medical university, Chongqing
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University; Pediatric Rheumatology division, Guangzhou
  - The Children's Hospibal ZheJiang University School of Medicine, Hangzhou
  - Chilren's hospital of nanjing medical university; Rheumatoid immunology, Nanjing
  - Shanghai Children's Medical Center; Renal rheumatology, Shanghai
  - Children's Hospital of Fudan University, Shanghai
  - The Second Affiliated Hospital & Yuying Children's Hospital of Wenzhou Medical College, Wenzhou